CLINICAL TRIAL: NCT02952885
Title: Strict IGF-1 Control in Acromegaly (I-Con Study)
Brief Title: Strict IGF-1 Control in Acromegaly
Acronym: I-Con
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCHIK-01
Record Dates: First submitted 2016-10-26; First posted 2016-11-02 (Estimated); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly | interventions — pegvisomant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pegvisomant (Experimental): Open-label, non-randomized single arm variable dose study of pegvisomant conducted in a real world setting.
  Interventions: Drug: Pegvisomant

INTERVENTIONS:
Drug: Pegvisomant — Study medications will be prescribed as per clinical practice with PEGV being added, or optimally dosed, at the Month 0 visit. Subjects who are naïve to PEGV should start their injections from 10 mg twice a week to 10 mg daily if used as combination therapy or 10 to 20 mg daily if used as monotherapy. Maximum dosing should not exceed 40mg/day. Dosing of PEGV can be adjusted as per clinical judgement to meet the normalization of IGF-1 levels (<1.0 ULN) in increments of 5-10mg/day. In the event of a reduction in IGF-1 below the LLN, the dose of PEGV could be decreased by 5-10 mg/day.
  Other Names: Somavert

SUMMARY:
Acromegaly is a rare, chronic, and debilitating disease, usually caused by a benign tumor on the pituitary gland, which leads to excessive production of growth hormone (GH). GH excess in turn causes overproduction of another hormone called insulin-like growth factor-1 (IGF-1). IGF-1 levels are currently the most widely accepted measure of disease activity.

In Canada, medical therapy with a type of medicine called "somatostatin analogues" (SSA), such as octreotide and lanreotide, is recommended for treatment of acromegaly. However, studies have shown that a significant number of patients who take SSA medications alone remain with elevated levels of IGF-1 in their blood.

Another medication that is used to treat acromegaly is pegvisomant (PEGV), and the investigators plan to study whether strict control of IGF-1, by adding or optimizing the use of PEGV, results in a significant health benefits to patients who still have modestly high levels of IGF-1 in their blood.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (at least 18 years old) with confirmed acromegaly whose IGF-I levels are persistently but modestly (1.0 ULN < [IGF-1 serum level] < 1.5 ULN) elevated following medical therapy such as SSA, PEGV, cabergoline alone or in combination.

Exclusion Criteria:

1. Progressive or recent visual field loss or optic chiasmal compression, or pituitary tumors within 2mm from the chiasm. Patients whose visual field loss, optic chiasmal compression or pituitary tumor has been stable for at least a year will be eligible.
2. Cranial nerve palsies or intracranial hypertension requiring tumour decompression surgery
3. Clinically significant hepatic disease and/or elevated liver enzymes (ALT, AST > 3 x ULN)
4. Patients who have received pituitary surgery within one year prior to screening visit
5. Patients who have received radiation therapy within one year prior to screening visit
6. History of hypersensitivity to any components of Pegvisomant
7. Inability to fully comprehend the nature of the study or cooperate with study procedures
8. Pregnant / lactating women and subjects refusing to use adequate contraception to prevent pregnancy during the study.
9. Subjects unwilling or unable to self-administer medication on a daily basis
10. known or suspected alcohol / drug abuse
11. Severe acute or chronic medical or psychiatric condition or laboratory abnormality that could increase the risk associated with trial participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-07-27 (Actual); Primary Completion 2020-05-07 (Actual); Study Completion 2020-05-07 (Actual)

PRIMARY OUTCOMES:
Health Related Quality of Life (AcroQoL) | six months

SECONDARY OUTCOMES:
Serum IGF-1 level | six months
Acromegaly Disease Activity Tool (ACRODAT) | six months
  To assess acromegaly co-morbidities
Patient-assessed Acromegaly Symptom Questionnaire | six months
  To assess acromegaly signs and symptoms
Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment | six months

CONTACTS AND LOCATIONS:
Overall Officials: Constance Chik, MD, Principal Investigator — St. Michael's Hospital, Toronto, ON
Locations (5):
- Canada (5):
  - University of Alberta Hospital, Edmonton, Alberta
  - St. Joseph Health Care London, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - McGill University Health Centre, Montreal, Quebec
  - Centre hospitalier universitaire de Québec-Université Laval, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No